CLINICAL TRIAL: NCT01136200
Title: Impact of Infectious Diseases Specialists on the Appropriateness of Antimicrobial Therapy in Surgical and Medical Wards: a Multicenter Randomized Controlled Trial.
Brief Title: Impact of Infectious Diseases Specialists on the Appropriateness of Antimicrobial Therapy in Surgical and Medical Wards
Acronym: ATBREFSURMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Philippe LESPRIT, Dr Philippe LESPRIT, Henri Mondor University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREQHOS 08023
Record Dates: First submitted 2010-05-28; First posted 2010-06-03 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Patients Receiving Antimicrobial Therapy
Keywords: Surgical and medical wards; Adults; Antimicrobial therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infectious disease specialist advice (Experimental): Patients receiving the intervention (infectious disease specialist advice)
  Interventions: Other: Infectious disease specialist advice
- Control (No Intervention): Patients not receiving infectious disease specialist advice

INTERVENTIONS:
Other: Infectious disease specialist advice — Indication, choice, dosing and duration of antimicrobial therapy
  Arms: Infectious disease specialist advice

SUMMARY:
CONTEXT: Antibiotics are frequently used in hospital but the appropriateness of prescriptions ranged between 25-50%. The intervention of infectious disease specialists (IDS) could improve the appropriateness of prescriptions and reduce their use. The impact of IDS has not been yet fully estimated using a randomized trial to compare the quality of care of patients who will benefit of the intervention.

OBJECTIVES: To show using a randomized trial that patients with IDS advice will receive more appropriate antimicrobial therapy but less exposure to antibiotics, as compared to patients who will not receive IDS advice.

METHODS: Prospective randomized trial comparing antibiotic exposure and appropriateness of prescriptions in two groups of patients:

* Control group: antibiotic prescriptions will be initiated and managed by the attending physicians
* Intervention group: antibiotic prescriptions will be systematically evaluated by the IDS and changed if judged necessary by the attending physicians, following IDS' advice.

STUDY PROCESS: The study will took place in 4 university hospitals. Two medical or surgical wards will participate by hospital. For each ward, the period of the study will be 2 x 4 weeks.Total duration of the study: 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Hospitalized in surgical or medical wards
* Receiving antimicrobial therapy for active infection or prolonged surgical prophylaxis
* Therapy prescribed by the attending ward physician

Exclusion Criteria:

* Patients receiving antimicrobial therapy not prescribed by the attending ward physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Appropriateness of antimicrobial therapy | Between days 7 and 10 after starting antimicrobial therapy
  Appropriateness of antimicrobial therapy will be evaluated at the start, between days 3 and 5, and at the end of therapy (between days 7 and 10).

SECONDARY OUTCOMES:
Clinical impact | Between days 7 and 10 after starting antimicrobial therapy
  Length of hospitalization;clinical outcome: resolution of infection; in hospital mortality
Antibiotic exposure | 14 days
  Antibiotic exposure will be evaluated using the following parameters:
  number of days of therapy/numbers of days of hospitalization; defined daily doses of antibiotic/number of days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lesprit, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor University Hospital, Créteil, France

REFERENCES:
- [Derived] Lesprit P, de Pontfarcy A, Esposito-Farese M, Ferrand H, Mainardi JL, Lafaurie M, Parize P, Rioux C, Tubach F, Lucet JC. Postprescription review improves in-hospital antibiotic use: a multicenter randomized controlled trial. Clin Microbiol Infect. 2015 Feb;21(2):180.e1-7. doi: 10.1016/j.cmi.2014.08.015. Epub 2014 Oct 14. PMID 25658564